CLINICAL TRIAL: NCT02489487
Title: Phase I, Drug-drug Interaction Study in Healthy Volunteers to Investigate the Safety, Tolerability and Pharmacokinetics of VM-1500 When Administered Orally, in Combination With Raltegravir or Darunavir
Brief Title: Study in Healthy Volunteers to Investigate the Safety, Tolerability and Pharmacokinetics of VM-1500
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VM-1500-002
Record Dates: First submitted 2015-06-18; First posted 2015-07-03 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: HIV-infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- VM-1500 + Raltegravir (Experimental): VM-1500 40 mg in combination with 400 mg Raltegravir
  Interventions: Drug: VM-1500; Drug: Raltegravir
- VM-1500 +Darunavir (Experimental): VM-1500 40 mg in combination with 600 mg Darunavir boosted with 100 mg Ritonavir
  Interventions: Drug: VM-1500; Drug: Darunavir; Drug: Ritonavir
- VM-1500 (Experimental): VM-1500 40 mg alone
  Interventions: Drug: VM-1500

INTERVENTIONS:
Drug: VM-1500 — VM-1500 40 mg
Drug: Darunavir — Darunavir 600 mg
  Arms: VM-1500 +Darunavir
Drug: Ritonavir — Ritonavir 100 mg
  Arms: VM-1500 +Darunavir
Drug: Raltegravir — 400 mg Raltegravir
  Arms: VM-1500 + Raltegravir

SUMMARY:
A randomized single dose, drug-drug interaction study in healthy volunteers for VM - 1500 given alone or in combination with Raltegravir or Darunavir in a 3 arm approach. The parallel design is used due to the long half life for VM-1500.

DETAILED DESCRIPTION:
This drug-drug interaction study will not be done as a cross-over study due to the extreme long half life of the drug. The 24 healthy subjects participating will be randomized to VM-1500 alone or VM-1500 in combination with Raltegravir or Darunavir in parallel arms.

For the cohort taking VM-1500 40 mg only just 4 subject will be enrolled as 6 subjects have been already on the same regimen in the trial before. Based on the parallel design it seems appropriate not to expose more healthy subjects than necessary. This means the available data of 6 subjects dosed with 40 mg VM-1500 alone will be matched.

Three groups of healthy subjects will be randomized to VM-1500 alone or VM-1500 in combination with Raltegravir or Darunavir (4:10:10). The healthy subjects will stay at the unit and receive 40 mg VM-1500 alone or VM1500 in combination with Raltegravir or Darunavir one time and PK blood samples at several time points will be collected. PK (trough level) blood samples will also be collected at visits on Days 2, 4,7, 14, 21, and on Day 36.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects age between 18-45 years
2. Has been determined healthy by physical examination, assessment of drug abuse, medical history and vital signs
3. Has normal or acceptable results for the following screening tests: complete blood count (CBC), blood urea nitrogen (BUN), serum creatinine (Cr), fasting blood sugar (FBS), total bilirubin, aspartate aminotransferase (AST or SGOT), alanine aminotransferase (ALT or SGPT), alkaline phosphatase (ALP) and urinalysis.
4. Negative result for hepatitis A, hepatitis B, hepatitis C and HIV antibodies
5. Willing to participate and signed the informed consent form

Exclusion Criteria:

1. Hepatic or kidney disorders or any other disease or disorder which may in the opinion of the Investigator interfere with the results of the study or threaten the health of volunteers;
2. Drug intake (including herbal drugs) during the last month;
3. Active alcohol and/or drug abuse that, in the opinion of the site investigator, would interfere with adherence to study requirements;
4. Volunteers have taken any investigational drug at least 3 month prior to the start of the study;
5. Inability to understand the Protocol or follow its instructions.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Division of AIDS table for grading the severity of ADULT Adverse Events | 36 days
  Safety and tolerability of VM-1500 alone or in combination with raltegravir or darunavir in adult healthy subjects

SECONDARY OUTCOMES:
Plasma concentrations of VM-1500 from Day 1 to Day 36 | 36 days
  Plasma concentrations of VM-1500 given alone or in combination with raltegravir or darunavir
Plasma concentrations of VM1500A (active metabolite of VM1500) from Day 1 to Day 36 | 36 days
  Plasma concentrations of VM-1500A alone or in combination with raltegravir or darunavir

CONTACTS AND LOCATIONS:
Overall Officials: Somruedee Chatsiricharoenkul, MD, Principal Investigator — Acriles
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Bangkok, Wanglang Road, Thailand

IPD SHARING:
Plan to Share IPD: No